CLINICAL TRIAL: NCT04915066
Title: Probability and Factors Associated With Early Discontinuation of Insulin Pump Therapy in Adults With Diabetes at the Center Hospitalier Sud Francilien
Brief Title: Study of Insulin Pump Discontinuation in Adults With Diabetes
Acronym: STOPPOMPE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0012
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus, type 1; Diabetes mellitus, type 2; Insulin Infusion Systems; Patient Education
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical data collection — Collection of medical data from patients'medical records

SUMMARY:
The purpose of this study is to determine the rate of insulin pump discontinuation 18 months after initiation in patients with diabetes, and to determine factors associated with this discontinuation.

DETAILED DESCRIPTION:
Insulin pump discontinuation has been mostly studied in children and young adults living with diabetes, and rarely with a time-to-event analysis. We aim to evaluate the rate of insulin pump discontinuation after 18 months from initiation and factors associated with it in adults with diabetes.

Knowing these factors would allow better support for patients in difficulty.

ELIGIBILITY:
Inclusion Criteria:

All patients (adults and adolescents) with diabetes and an insulin pump initiation from 1 January 2015 to 30 June 2018 in the diabetes department of the Centre hospitalier sud francilien.

Exclusion Criteria:

* Pregnant women (or women planning pregnancy in the short term) with an insulin pump initiation from 1 January 2015 to 30 June 2018
* Patients hospitalized for an insulin pump replacement or change between 1 January 2015 and 30 June 2018.
* Patients with a history of insulin pump initiation within a period of less than 6 months before a new pump start between 1 January 2015 and 30 June 2018.

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Sample of patients from the diabetes department of a public hospital in France (Corbeil-Essonnes).
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Permanent discontinuation of insulin pump use. | at 18 months
  Insulin pump discontinuation is considered permanent if > 6 consecutive months with patient back to insulin pen and no use of pump-related consumables during the 6 months.

SECONDARY OUTCOMES:
Age | at day 0
  Age of patient at the moment of insulin pump discontinuation.
Sex | at day 0
  Sex of patient
type of diabete | at day 0
  type 1 or 2

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No